CLINICAL TRIAL: NCT02380729
Title: Mutation Exploration in Non-acquired, Genetic Disorders and Its Impact on Health Economy and Life Quality
Acronym: MENDEL
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Markus Schuelke, M.D., Professor, Charite University, Berlin, Germany
Other Study IDs: EA2_107_14
Record Dates: First submitted 2015-02-18; First posted 2015-03-05 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Genetic Diseases
Keywords: Health care delivery; Human Phenotype Ontology; Mutation prioritization; Next Generation Sequencing; Mutation detection; Bioinformatic analysis; Quality of life
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — Whole Genome Sequencing

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from peripheral blood cells of the index patient and of his/her parents.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Index patients: Children between birth and 18 years of age manifesting with a suspected genetic disorder.
  Investigation: First Gene Panel Sequencing and if no mutation ist found > Whole Genome Sequencing (WGS)
  Interventions: Genetic: Gene Panel Sequencing; Genetic: Whole Genome Sequencing (WGS)
- Parents of the index patient: Both parents of the index patient.
  Investigation: Whole Genome Sequencing (WGS) if no mutation is found by Gene Panel Sequencing of the index patient.
  Interventions: Genetic: Whole Genome Sequencing (WGS)

INTERVENTIONS:
Genetic: Gene Panel Sequencing — Enrichment for and panel sequencing of 2942 disease genes listed in the Online Mendelian Inheritance of Man (OMIM) database.
  Groups: Index patients
Genetic: Whole Genome Sequencing (WGS) — Whole Genome Sequencing of the index case and of both parents in the event that Gene Panel Sequencing did not identify a disease-causing mutation.

SUMMARY:
The MENDEL-study will investigate whether the use of gene panel or whole genome sequencing (WGS) will:

1. improve the rate of diagnosis and through this compare the performance of the two diagnostic approaches (gene panel vs. WGS),
2. investigate whether use of said sequencing approaches early in the diagnostic process results in reduced health care spending, and
3. result in an improved quality of life for the patients and their parents.

DETAILED DESCRIPTION:
Patients will be recruited from in- and outpatient clinics at the Otto Heubner Center, the Berlin Center for Rare Diseases, and the Institute for Medical Genetics and Human Genetics at Charité-Universitätsmedizin Berlin, Germany. Following informed consent, 5 ml EDTA blood will be obtained from the index case and 10 ml blood from each parent. Disease related phenotype information and the outcome of previous diagnostic tests and procedures will be recorded as part of Study visit #1.

[1] Study visit #1

1. A medical genetics physical will be performed. Detailed clinical symptoms (phenotype) will be recorded using Human Phenotype Ontology (HPO) terminology.
2. A detailed pedigree will be drawn.
3. Age of disease onset will be determined.
4. Results from previous diagnostic tests and procedures, as well as hospital stays, will be recorded.
5. The parents will be asked to complete a validated, standardized quality of life questionnaire adapted for for rare disease. The questionnaire is available online or in paper form.

[2] Study visit #2a (optional)

This study visit will only take place in the event that gene panel sequencing identifies a variant of uncertain significance, where additional information would be needed in order to determine its pathogenicity (e.g. confirmational biochemical testing, collection of additional information). Relevant research findings will be discussed and the nature and necessity of the additional testing will be explained.

[3] Study visit #2b (optional)

This study visit will only take place in the event that WGS identifies a variant of uncertain significance where additional information is needed in order to determine its pathogenicity > see Study visit #2a.

[4] Study visit #3 (results session)

Results will be returned in the context of a genetic counseling session.

[5] Study visit #4 (6 months after Study visit #3)

The parents will be asked to complete the validated, standardized quality of life questionnaire adapted for rare disease again.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: Suspicion of genetic disease. (Only one of the following criteria is required.) [1.1] Family member(s) with similar phenotype OR [1.2] At least two affected organ systems OR [1.3] One affected organ system that is known to be associated with multiple disease causing genes (e.g. long QT syndrome) OR [1.4] Multiple birth defects
2. Both parents must be available for blood draw in order to confirm phase (segregation analysis) or in order to perform WGS of the trio at a later time point.
3. Age: from birth up until age 18 years
4. Gender: Both sexes will be included

Exclusion Criteria:

1. Suspicion that the phenotype is due to an acquired disease
2. Missing informed consent from both parents or from all legal guardians for genetic testing in the setting of a clinical trial.
3. Clinical diagnosis of a disease with a known monogenic cause, e.g. Phenylketonuria or Cystic fibrosis.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Index patients: Children (age newborn to 18 years) who present with a suspected genetic disorder
  Parents: biological mother and father of each index case.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-01-31 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield through gene panel sequencing of 3089 known disease genes. | 6 months.
  The number of confirmed disease causing mutations that can be identified in 200 patients following gene panel sequencing and analysis with the PhenIX software.

SECONDARY OUTCOMES:
Quality of Life | 2 years
  Assessment of the parents' quality of life before and after molecular diagnostics and reception of a molecular genetic diagnosis.
Manageability of a next generation sequencing (NGS) pipeline in routine clinical diagnostics | 2 years
  Calculation of the duration [months] between recruitment of a family and the final genetic counselling.
Health economy of NGS | 2 years
  Comparison of the cost of "standard diagnostics" versus the use of gene panel sequencing or WGS at an early stage in the diagnostic process. Health economic analysis of the costs incurred for each patient through "the standard diagnostic approach" in comparison to costs incurred through the use of gene panel sequencing/WGS.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schuelke, M.D., Principal Investigator — Department of Neuropediatrics, Charité; Stefan Mundlos, M.D., Principal Investigator — Institute of Medical Genetics and of Human Genetics, Charité; Heiko Krude, M.D., Principal Investigator — Department of General Pediatrics, Charité
Locations (3):
- Germany (3):
  - Department of General Pediatrics, Charité-Universitätsmedizin, Berlin
  - Department of Neuropediatrics, Charité-Universitätsmedizin, Berlin
  - Institute of Medical Genetics and Human Genetics, Charité-Universitätsmedizin, Berlin

REFERENCES:
- [Background] Zemojtel T, Kohler S, Mackenroth L, Jager M, Hecht J, Krawitz P, Graul-Neumann L, Doelken S, Ehmke N, Spielmann M, Oien NC, Schweiger MR, Kruger U, Frommer G, Fischer B, Kornak U, Flottmann R, Ardeshirdavani A, Moreau Y, Lewis SE, Haendel M, Smedley D, Horn D, Mundlos S, Robinson PN. Effective diagnosis of genetic disease by computational phenotype analysis of the disease-associated genome. Sci Transl Med. 2014 Sep 3;6(252):252ra123. doi: 10.1126/scitranslmed.3009262. PMID 25186178